CLINICAL TRIAL: NCT00111956
Title: Effects of Tumor Necrosis Factor (TNF)-Alpha Antagonism in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNF-alpha (completed); F32DK068902 (NIH)
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Syndrome X
Keywords: TNF; metabolic syndrome; inflammation; CRP; adiponectin
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept
  Arms: Etanercept
Drug: Placebo
  Arms: Placebo

SUMMARY:
Metabolic syndrome is associated with increased inflammatory cytokines and reduced adiponectin, that may be mediated in part by TNF production from abdominal fat. We reasoned that an anti-TNF agent would reduce C-reactive protein (CRP) and increase adiponectin, improving the inflammatory milieu associated with metabolic syndrome.

DETAILED DESCRIPTION:
Screening visit 1:

Fifty six patients will be randomized to receive etanercept or identical placebo. During the screening visit, after informed consent is obtained, subjects will undergo a medical history and physical exam, which will include vital signs, weight, abdominal girth measurements and an evaluation for signs of underlying infection. A purified protein derivative (PPD) of 5 tuberculin units (TU) (0.1 milliliter of 5 TU/0.1 ml solution) will be intradermally placed to test for the presence of tuberculosis (TB). Fasting blood work will include a complete blood count (CBC), glucose, insulin, a cholesterol panel, and urine pregnancy test. Subjects will be shown what a subcutaneous injection entails using placebo. Patients will be selected based on their laboratory results, abdominal girth measurements and PPD negativity 48 hrs after placement.

Screening visit 2:

Subjects will return 48 hours after their first screening visit for evaluation of their PPD test. In the event of a positive PPD, subjects will be excluded from the study, and their primary care physicians will be notified of their test result.

Day 1 visit:

Subjects will report to Massachusetts General Hospital (MGH) or Massachusetts Institute of Technology (MIT) Clinical Research Center (GCRC) after an overnight fast. Fasting blood work will be obtained to test for CRP, adiponectin, IL-6, TNF-alpha, TNF-alpha receptor 1, TNF-alpha receptor 2, free fatty acids, glucose, insulin and a cholesterol panel, and CBC. A urine pregnancy test will be done. Patients will be asked to recall the food they consumed over the past 24 hours. A bionutritionist will measure height, weight, waist, hip, chest, arm, neck and thigh circumference. Subjects will be instructed to practice adequate birth control throughout the study. Serum will be stored for etanercept antibody testing.

Subjects will then undergo an insulin modified frequently sampled intravenous (IV) glucose tolerance test (FSIGT) as initially developed by Bergman et al.

Dual energy x-ray absorptiometry (DEXA) (Hologic QDR 4500) will be used to determine whole body and regional fat. The technique has a precision error (1 SD) of 3% for whole body fat and 1.5% for lean mass. Subjects will also undergo a single thin-slice CT scan of the abdomen at L4 vertebral body to determine visceral and subcutaneous fat area.

Indirect calorimetry for the measurement of resting energy expenditure indirect calorimetry using the Deltatrac instrument (Sensormedics, Anaheim, CA) will be carried out.

Drug administration:

Patients will be given a total of either etanercept 50 mg subcutaneously or placebo subcutaneously at the GCRC at the end of their visit. They will receive this in two injections of 25 mg each, one given immediately following the other, at different body sites. Etanercept will be supplied as a sterile, white, preservative-free, lyophilized powder. The pharmacy will reconstitute it with 1 mL of the supplied sterile bacteriostatic water for injection (BWFI), United States Pharmacopeia (USP) (containing 0.9% benzyl alcohol). Each vial of etanercept contains 25 mg etanercept, 40 mg mannitol, 10 mg sucrose, and 1.2 mg tromethamine. Subjects will receive the 50 mg dose of etanercept or placebo once a week, given as two 25 mg injections, one immediately following the other, at different body sites, at each of their ensuing three visits to the GCRC, on Visit Day 8, Visit Day 15 and Visit Day 22. Subjects will be monitored for 30 minutes after the injection of study drug at each visit. The skin injection site will be observed and their vital signs will be taken. If a subject has a significant exposure to varicella virus during the study, transient termination of the study will be considered.

Day 8 visit, Day 15 visit, Day 22 visit:

Subjects will report to MGH or MIT Clinical Research Center after an overnight fast. Each subject will undergo a history and physical exam to assess for safety and compliance. Fasting blood work will be obtained. A bionutritionist will measure subjects' height, weight, hip and waist circumference and calculate a waist to hip ratio. They will receive 50 mg of either etanercept or placebo, given as two 25 mg doses subcutaneously, at different body sites.

Day 25 visit:

Subjects will report to MGH or MIT Clinical Research Center after an overnight fast. Each subject will undergo a history and physical exam to assess for safety and compliance. Blood work, a urine pregnancy test and 24 hour food recall will be collected, identical to that on Day 1 visit. Anthropomorphic measurements will be the same as the Day 1 visit. Subjects will undergo an intravenous glucose tolerance test (IVGTT) identical to that on the Day 1 visit. Subjects will undergo a DEXA, bioelectric impedance analysis (BIA), and CT, and indirect calorimetry identical to those on the Day 1 visit. No study drug will be administered at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Hyperinsulinemia in the upper quartile of the non-diabetic population defined as ≥10 mU/mL (Framingham Data, oral communication, James Meigs, MD) or fasting glucose 110-126 mg/dL, plus two of the following: *Abdominal obesity defined by waist hip ratio > 0.90 for men and > 0.85 for women or *body mass index (BMI) > 30 kg/m2
* Dyslipidemia including serum triglycerides ≥150 mg/dl or serum HDL < 0.9 mmol/L for men (35 mg/dL) and < 1.0 mmol/L (39 mg/dL) for women
* Hypertension defined as blood pressure ≥ 140/90 or on medication

Exclusion Criteria:

* Positive PPD (≥ 5mm induration) on screening
* Current infection
* Therapy with glucocorticoid or immunosuppressant at time of recruitment or within past 3 months
* Reception of live vaccine within 1 week of recruitment
* History of blood dyscrasia including any kind of anemia, thrombocytopenia, pancytopenia. Women with a reversible cause of anemia that has resolved will be eligible.
* History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers who will be eligible)
* History of organ transplantation
* History of central nervous system (CNS) demyelinating disorder or any first degree relative with multiple sclerosis
* History of congestive heart failure (CHF) classes I-IV
* Current use of insulin, any oral anti-hyperglycemic agents, pentoxyfylline, beta-agonists
* Current use of fibrate or niacin
* Initiation of statin therapy within prior 6 weeks or expecting a change in statin dose over the upcoming 3 months
* Hemoglobin < 11 g/dl
* Positive pregnancy test
* Women of child-bearing potential not currently using non-hormonal birth control methods including barrier methods (intrauterine device (IUD), condoms, diaphragms) or abstinence
* Patients with known autoimmune or inflammatory conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP), mg/L | 25 days

SECONDARY OUTCOMES:
Adiponectin, ug/mL | 25 days
Interleukin 6, ng/L | 25 days
Fibrinogen, mg/dL | 25 days
Insulin sensitivity | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Bernstein LE, Berry J, Kim S, Canavan B, Grinspoon SK. Effects of etanercept in patients with the metabolic syndrome. Arch Intern Med. 2006 Apr 24;166(8):902-8. doi: 10.1001/archinte.166.8.902. PMID 16636217